CLINICAL TRIAL: NCT03718832
Title: Fresh Food Farmacy: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John B Bulger, DO (Other)
Collaborators: Massachusetts Institute of Technology (Other); Cornell University (Other); Stanford University (Other); Geisinger Clinic (Other)
Responsible Party: Sponsor-Investigator, John B Bulger, DO, Chief Health Officer, GIO, Geisinger Clinic
Organization: Geisinger Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-0297
Record Dates: First submitted 2018-10-17; First posted 2018-10-25 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group-Begin Now (Experimental): Group 1- Will be randomized to the treatment ("Begin Now") group for the Fresh Food Farmacy program. Subjects will be consented to join the FFF study prior to learning their program start date. They will join the FFF program right away when the program opens in their geographic area. Data will be collected during the first 12 months of subject participation and EHR and claims data may be analyzed for an additional 12 month follow-up period (24 months in total).
  Interventions: Other: Fresh Food Farmacy
- Control Group-Begin Later (No Intervention): Group 2- Will be randomized to the control ("Begin Later") group for the FFF program. These subjects will be consented to join the FFF study prior to learning their program start date. They will join the FFF program approximately 6 months after the program opens in their geographic area. Data will be collected during the first 6 months of subject participation and used as control data for the study. EHR and claims data may be analyzed for an additional 12 month follow-up period (24 months in total from the start of the trial).

INTERVENTIONS:
Other: Fresh Food Farmacy — Patients are prescribed fresh food by a dietician, fill the prescription each week at the FFF clinic, receive training on how to use the food, and training in diabetes self management.
  Arms: Treatment Group-Begin Now

SUMMARY:
This trial investigates the value created by the highly innovative Fresh Food Farmacy (FFF) program at Geisinger Health. The program provides food-insecure diabetics with healthy food for their entire household: at least two meals per day, five days a week. The program also provides education on how to prepare the food, and education on healthy living including diabetes self management. The research measures the effects of the FFF program on patient health and wellbeing.

DETAILED DESCRIPTION:
This is a pragmatic, prospective, randomized controlled trial of Geisinger's Fresh Food Farmacy (FFF) program as the program expands to new sites. Qualifying subjects will be randomized 1:1 to receive either early participation in the FFF program (treatment group) or later participation (control group).

Approximately 500 Geisinger subjects will participate in this study with about half assigned to the treatment group and about half to the control group. The treatment group will begin the program soon after trial recruitment: the "Begin Now" group. The control group will begin the program after 6 months: the "Begin Later" group. Approximately 2000 household members will be included in the data-only portion of the research.

Outcomes will include clinical measures, such as HbA1c, survey responses including self-assessed health measures, and utilization / healthy-behavior measures from EHR and paid claims data. These will be measured for subjects and their household members.

ELIGIBILITY:
Inclusion Criteria:

* Type II Diabetes and an HbA1c ≥ 8.0 as determined by the most recent measurement in the Geisinger EMR within the prior 12 months
* Food insecure based on a two-question survey instrument
* Age > 17 & Age <86
* Living within geographic reach of the program (Lewistown, PA and Scranton, PA)

Exclusion Criteria:

* Already enrolled in FFF in Shamokin
* Not English speaking (working on changing this as the program evolves)
* On hospice or palliative care
* Acute or chronic psychosis
* Resides in a facility which provides meals
* Active medical disorder that would preclude participation in the classes, weekly clinic visits, or result in a limited diet, including:

  * Cancer; active treatment
  * Steroid dependent asthma/ COPD/ emphysema
  * Steroid dependent Colitis
  * Chronic Kidney Disease with GFR< 30 mg/mmol
  * Celiac disease
  * Cirrhosis
  * Steroid dependent arthritis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Bulger, MD, Principal Investigator — Geisinger Clinic; Joseph J Doyle, Principal Investigator — MIT Sloan School of Management
Locations (2):
- United States (2):
  - Fresh Food Farmacy, Lewistown, Pennsylvania
  - Fresh Food Farmacy, Scranton, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data at the subject level, pending approval from the IRB and Geisinger.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Available pending approval from the IRB and after primary publication.
Access Criteria: To be determined

REFERENCES:
- [Background] Doyle J, Alsan M, Skelley N, Lu Y, Cawley J. Effect of an Intensive Food-as-Medicine Program on Health and Health Care Use: A Randomized Clinical Trial. JAMA Intern Med. 2024 Feb 1;184(2):154-163. doi: 10.1001/jamainternmed.2023.6670. PMID 38147326
- Available data/document: Individual Participant Data Set: doi:10.7910/DVN/LZUTU0 — https://doi.org/10.7910/DVN/LZUTU0
- Available data/document: Analytic Code: doi:10.7910/DVN/LZUTU0 — https://doi.org/10.7910/DVN/LZUTU0

RESULTS

PARTICIPANT FLOW:
Period: Analysis Sample
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Started | 249 | 251
Completed | 230 | 235
Not Completed | 19 | 16
Not completed — Withdrawal by Subject | 18 | 15
Not completed — Legal hold on data | 1 | 0
Not completed — Participant from treated household | 0 | 1
Period: 6-month HbA1c Sample
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Started | 230 | 235
Completed | 170 | 179
Not Completed | 60 | 56
Not completed — Lost to Follow-up | 60 | 56

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later | Total
Number analyzed (Participants) | 230 | 235 | 465
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (11.3) | 54.4 (12.4) | 54.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 125 | 255
  Male | 100 | 110 | 210
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic (any race) | 16 | 23 | 39
  Non-Hispanic Black | 23 | 18 | 41
  Non-Hispanic White | 189 | 189 | 378
  Non-Hispanic and other race | 2 | 5 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 230 | 235 | 465
Prior-year healthcare use [Count of Participants; unit: Participants]
  Any inpatient admission | 59 | 48 | 107
  Any emergency department visit | 97 | 94 | 191
Clinic location [Count of Participants; unit: Participants]
  Rural | 64 | 67 | 131
  Urban | 166 | 168 | 334

OUTCOME MEASURES:

1. Primary Outcome: HbA1c
Description: Glycated hemoglobin (HbA1c) is a measure of the average share of glucose that has been in the bloodstream over the 2-3 months preceding measurement. HbA1c is measured by performing assays on samples of the participants' blood.
  Units are percentages; for differences between HbA1c values, units are percentage points.
  An HbA1c value of 6.5% is the lower threshold for type 2 diabetes. HbA1c values are rarely above 15-20%. In the context of this study (patients with type 2 diabetes), higher scores are considered a worse outcome.
Time Frame: 6 months after trial enrollment
Population: Participants from the 465-person analysis sample who completed an HbA1c blood test between 5 and 10 months after program enrollment.
Measure: Mean (Standard Deviation); unit: % of hemoglobin
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 170 | 179
% of hemoglobin | 8.781177 (1.643995) | 8.814526 (1.978937)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.8638688, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -0.0333487, 95% CI 2-sided [-0.415628 to 0.3489306], Standard Error of Mean 0.1943638
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.9714571, Regression, Linear — Adjusted mean difference for full prespecified controls; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -0.0066385, 95% CI 2-sided [-0.371329 to 0.358052], Standard Error of Mean 0.1853917

2. Secondary Outcome: HbA1c
Description: Glycated hemoglobin. Units are percentages (for differences, percentage points) reflecting the average share of glucose in the bloodstream over the previous 2-3 months.
  An HbA1c value of 6.5% is the lower threshold for type 2 diabetes. HbA1c values are rarely above 15-20%.
  In the context of this study (patients with type 2 diabetes), higher scores are considered a worse outcome.
Time Frame: 12 months after trial enrollment
Measure: Mean (Standard Deviation); unit: % of hemoglobin
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 164 | 161
% of hemoglobin | 8.735975 (1.748229) | 8.595031 (2.035983)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.5039565, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 0.1409446, 95% CI 2-sided [-0.2735162 to 0.5554053], Standard Error of Mean 0.2106711
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.5684854, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.1213915, 95% CI 2-sided [-0.2970052 to 0.5397882], Standard Error of Mean 0.2126328

3. Secondary Outcome: Fasting Glucose
Description: Fasting blood glucose is a measure of blood sugar control over a short time period (the blood glucose content after an overnight fast).
  Units are mg/dL. To convert to mmol/L (SI), multiply by 0.0113. Lower fasting blood glucose levels indicate better health within the context of this study.
Time Frame: 6 and 12 months after trial enrollment
Population: Number of participants analyzed differs due to differences in the number of participants who completed blood tests between 6 and 12 months after trial enrollment.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 127 | 137
mg/dL
  6 months after trial enrollment | 185.0236 (76.36467) | 198.292 (99.97935)
  12 months after trial enrollment: number analyzed (Participants) | 115 | 93
  12 months after trial enrollment | 185.4696 (68.86821) | 172.3441 (68.18301)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.2247426, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -13.26835, 95% CI 2-sided [-34.73804 to 8.201347], Standard Error of Mean 10.90353
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.2794015, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -12.20164, 95% CI 2-sided [-34.37119 to 9.9679], Standard Error of Mean 11.25555
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.1708328, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 13.12548, 95% CI 2-sided [-5.703702 to 31.95466], Standard Error of Mean 9.550462
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.2801138, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 11.47577, 95% CI 2-sided [-9.422762 to 32.3743], Standard Error of Mean 10.59479

4. Secondary Outcome: Weight (lb)
Description: Weight in pounds. In the context of this study, higher values are considered a worse outcome.
  SI conversion factor: To convert pounds to kilograms, multiply by 0.4536.
Time Frame: 6 and 12 months after trial enrollment
Population: Number of participants analyzed differs due to differences in the number of participants who had their weight recorded between 6 and 12 months after trial enrollment.
Measure: Mean (Standard Deviation); unit: pounds (lb)
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 195 | 205
pounds (lb)
  6 months after trial enrollment | 230.8205 (60.13527) | 238.9561 (66.3286)
  12 months after trial enrollment: number analyzed (Participants) | 181 | 187
  12 months after trial enrollment | 227.9171 (58.1217) | 237.5989 (63.47953)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.1991028, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -8.135585, 95% CI 2-sided [-20.57023 to 4.299061], Standard Error of Mean 6.325031
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.0480884, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 3.493798, 95% CI 2-sided [0.0295297 to 6.958066], Standard Error of Mean 1.761916
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.1276817, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -9.681804, 95% CI 2-sided [-22.15188 to 2.788269], Standard Error of Mean 6.34136
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.3318554, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 1.658257, 95% CI 2-sided [-1.698022 to 5.014535], Standard Error of Mean 1.706497

5. Secondary Outcome: Body Mass Index
Description: Body Mass Index (BMI) in kg/m^2. BMI is computed using weight (lb) and height (in). The CDC's healthy reference range for BMI among adults aged 20 and older is 18.5 to 24.9. BMI values greater than or equal to 30.0 indicate obesity. In the context of this study, higher BMI is considered a worse outcome.
Time Frame: 6 and 12 months after trial enrollment
Population: Number of participants analyzed differs due to differences in the number of participants whose weight was recorded between 6 and 12 months after trial enrollment.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 195 | 205
kg/m^2
  6 months after trial enrollment | 36.77117 (8.615884) | 37.6461 (10.06821)
  12 months after trial enrollment: number analyzed (Participants) | 181 | 187
  12 months after trial enrollment | 36.20175 (8.299285) | 37.65195 (9.895644)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.3502313, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -0.8749266, 95% CI 2-sided [-2.714084 to 0.9642311], Standard Error of Mean 0.9355095
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.0390797, Regression, Linear — Adjusted mean difference for full controls; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 0.5608222, 95% CI 2-sided [0.0282451 to 1.093399], Standard Error of Mean 0.2708671
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.1281032, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -1.450197, 95% CI 2-sided [-3.320109 to 0.419716], Standard Error of Mean 0.9508997
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.3044732, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.2794625, 95% CI 2-sided [-0.2549974 to 0.8139224], Standard Error of Mean 0.2717457

6. Secondary Outcome: Total Cholesterol
Description: Total cholesterol in mg/dL. The CDC recommends total cholesterol levels around 150 mg/dL and classifies levels of 200 mg/dL and above as unhealthy (hyperlipidemia). In the context of this study, higher total cholesterol indicates a worse outcome.
  SI conversion factor: To convert from mg/dL to mmol/L, multiply by 0.0259.
Time Frame: 6 and 12 months after trial enrollment
Population: Number of participants analyzed differs due to differences in the number of participants who completed blood tests including cholesterol measurements between 6 and 12 months after trial enrollment.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 149 | 161
mg/dL
  6 months after trial enrollment | 170.3087 (55.49542) | 160.5404 (48.39021)
  12 months after trial enrollment: number analyzed (Participants) | 145 | 134
  12 months after trial enrollment | 164.8345 (50.04346) | 165.3806 (56.96481)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.1007463, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 9.768353, 95% CI 2-sided [-1.907847 to 21.44455], Standard Error of Mean 5.933945
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.3859868, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 4.472004, 95% CI 2-sided [-5.66534 to 14.60935], Standard Error of Mean 5.150772
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.9324908, Regression, Linear — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -0.5461143, 95% CI 2-sided [-13.22545 to 12.13323], Standard Error of Mean 6.440905
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.6328075, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -2.752831, 95% CI 2-sided [-14.08487 to 8.579205], Standard Error of Mean 5.754947

7. Secondary Outcome: LDL Cholesterol
Description: Low-density lipoprotein (LDL) cholesterol, measured in mg/dL. The CDC recommends LDL levels of 100 mg/dL or below. In the context of this study, higher levels of LDL indicate a worse outcome.
  SI conversion factor: To convert from mg/dL to mmol/L, multiply by 0.0259.
Time Frame: 6 and 12 months after trial enrollment
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 151 | 158
mg/dL
  6 months after trial enrollment | 93.54835 (44.67019) | 85.19621 (36.72769)
  12 months after trial enrollment: number analyzed (Participants) | 142 | 131
  12 months after trial enrollment | 87.36268 (36.73616) | 84.72519 (36.62367)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.0743062, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 8.352141, 95% CI 2-sided [-0.8250086 to 17.52929], Standard Error of Mean 4.663846
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.1270654, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 5.971188, 95% CI 2-sided [-1.709219 to 13.65159], Standard Error of Mean 3.902349
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.553277, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 2.637485, 95% CI 2-sided [-6.110146 to 11.38512], Standard Error of Mean 4.443227
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.519562, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 2.53149, 95% CI 2-sided [-5.198658 to 10.26164], Standard Error of Mean 3.925307

8. Secondary Outcome: HDL Cholesterol
Description: High-density lipoprotein (HDL) cholesterol, measured in mg/dL. The CDC recommends HDL levels of at least 40 mg/dL in men and 50 mg/dL in women. In the context of this study, higher levels of HDL indicate a better outcome.
  SI conversion factor: To convert mg/dL to mmol/L, multiply by 0.0259.
Time Frame: 6 and 12 months after trial enrollment
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 149 | 161
mg/dL
  6 months after trial enrollment | 41.27718 (12.98269) | 41.8323 (12.08006)
  12 months after trial enrollment: number analyzed (Participants) | 144 | 135
  12 months after trial enrollment | 42.34722 (12.73743) | 43.73333 (17.07761)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.6976216, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -0.555117, 95% CI 2-sided [-3.363839 to 2.253605], Standard Error of Mean 1.427417
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.6329035, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -0.4977997, 95% CI 2-sided [-2.546815 to 1.551216], Standard Error of Mean 1.041102
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.445181, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -1.386111, 95% CI 2-sided [-4.954999 to 2.182777], Standard Error of Mean 1.812939
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.5542241, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -1.101914, 95% CI 2-sided [-4.765783 to 2.561956], Standard Error of Mean 1.860687

9. Secondary Outcome: Triglycerides
Description: Triglycerides, measured in mg/dL. The CDC recommends levels of triglycerides below 150 mg/dL. In the context of this study, higher levels of triglycerides indicate worse outcomes.
  SI conversion factor: To convert mg/dL to mmol/L, multiply by 0.0113.
Time Frame: 6 and 12 months after trial enrollment
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 149 | 162
mg/dL
  6 months after trial enrollment | 223.5705 (155.5674) | 201.0123 (157.1144)
  12 months after trial enrollment: number analyzed (Participants) | 143 | 132
  12 months after trial enrollment | 212.7762 (153.4214) | 224.1288 (268.9378)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.2045348, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 22.55812, 95% CI 2-sided [-12.35316 to 57.4694], Standard Error of Mean 17.74244
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.3675252, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 13.49781, 95% CI 2-sided [-15.93658 to 42.9322], Standard Error of Mean 14.95579
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.6709307, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -11.35256, 95% CI 2-sided [-63.8992 to 41.19407], Standard Error of Mean 26.69115
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.6766844, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -8.912496, 95% CI 2-sided [-50.95358 to 33.12859], Standard Error of Mean 21.34891

10. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure, measured in mm Hg. The CDC identifies normal healthy systolic blood pressure as below 120 mm Hg. The American College of Cardiology identifies 120 to 129 mm Hg as elevated blood pressure and 130 mm Hg and higher as hypertensive. Higher systolic blood pressure levels indicate worse outcomes.
Time Frame: 6 and 12 months after trial enrollment
Population: Number of participants analyzed differs due to differences in the number of participants who had their blood pressure recorded between 6 and 12 months after trial enrollment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 186 | 192
mm Hg
  6 months after trial enrollment | 128.3118 (19.06545) | 130.1823 (20.29064)
  12 months after trial enrollment: number analyzed (Participants) | 170 | 181
  12 months after trial enrollment | 126.0235 (17.24071) | 129.7956 (18.45165)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.356123, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -1.870464, 95% CI 2-sided [-5.851219 to 2.110291], Standard Error of Mean 2.024497
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.6566494, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -0.8636408, 95% CI 2-sided [-4.681041 to 2.95376], Standard Error of Mean 1.941141
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.0484944, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -3.772051, 95% CI 2-sided [-7.519021 to -0.0250809], Standard Error of Mean 1.905125
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.234947, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -2.167034, 95% CI 2-sided [-5.749627 to 1.415558], Standard Error of Mean 1.821244

11. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure, measured in mm Hg. The American College of Cardiology identifies normal diastolic blood pressure as below 80 mm Hg and elevated/hypertensive diastolic blood pressure as 80 mm Hg or above. Higher levels of diastolic blood pressure indicate worse outcomes.
Time Frame: 6 and 12 months after trial enrollment
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 186 | 192
mm Hg
  6 months after trial enrollment | 74.2043 (10.71504) | 74.76041 (10.40413)
  12 months after trial enrollment: number analyzed (Participants) | 170 | 181
  12 months after trial enrollment | 74.48235 (9.271847) | 73.98343 (10.46395)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.6091477, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -0.5561156, 95% CI 2-sided [-2.693002 to 1.58077], Standard Error of Mean 1.086759
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.713942, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -0.3787962, 95% CI 2-sided [-2.409379 to 1.651786], Standard Error of Mean 1.032547
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.6362064, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 0.4989275, 95% CI 2-sided [-1.573807 to 2.571662], Standard Error of Mean 1.053869
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.2748884, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 1.146286, 95% CI 2-sided [-0.9154561 to 3.208027], Standard Error of Mean 1.048105

12. Secondary Outcome: Times Eating Fruit in the Past 7 Days
Description: Patient-reported measure of diet improvement: Number of times in the last 7 days when the patient ate fruit.
Time Frame: 6 and 12 months after trial enrollment
Population: Number of participants analyzed differs due to differences in survey (non)response between surveys completed at 6 and 12 months after trial enrollment.
Measure: Mean (Standard Deviation); unit: # times
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 163 | 170
# times
  6 months after trial enrollment | 5.564417 (3.344494) | 5.241177 (3.397799)
  12 months after trial enrollment: number analyzed (Participants) | 144 | 137
  12 months after trial enrollment | 5.097222 (2.377986) | 5.79562 (3.343428)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.3823224, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 0.3232407, 95% CI 2-sided [-0.4036366 to 1.050118], Standard Error of Mean 0.3695066
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.4829339, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.2619965, 95% CI 2-sided [-0.4718566 to 0.9958495], Standard Error of Mean 0.3729922
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.045506, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -0.6983982, 95% CI 2-sided [-1.382737 to -0.0140597], Standard Error of Mean 0.3476441
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.0625551, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -0.6239824, 95% CI 2-sided [-1.280906 to 0.0329412], Standard Error of Mean 0.3336405

13. Secondary Outcome: Times Eating Dark Green Vegetables in the Past 7 Days
Description: Patient-reported measure of diet improvement: Number of times in the last 7 days when the patient ate dark green vegetables.
Time Frame: 6 and 12 months after trial enrollment
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: # times
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 163 | 170
# times
  6 months after trial enrollment | 6.288343 (20.69643) | 4.011765 (2.9007)
  12 months after trial enrollment: number analyzed (Participants) | 143 | 138
  12 months after trial enrollment | 4.202797 (2.378186) | 5.782609 (8.36899)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.1650343, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 2.276579, 95% CI 2-sided [-0.9420086 to 5.495166], Standard Error of Mean 1.636162
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.1442126, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 1.989458, 95% CI 2-sided [-0.6843682 to 4.663284], Standard Error of Mean 1.359013
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.0335498, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -1.579811, 95% CI 2-sided [-3.03574 to -0.1238828], Standard Error of Mean 0.739612
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.0398937, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -1.764632, 95% CI 2-sided [-3.447175 to -0.0820899], Standard Error of Mean 0.8545352

14. Secondary Outcome: Times Drinking Sweetened Beverages in the Past 7 Days
Description: Patient-reported measure of diet improvement: Number of times in the last 7 days when the patient drank sweetened beverages.
Time Frame: 6 and 12 months after trial enrollment
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: # times
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 162 | 167
# times
  6 months after trial enrollment | 2.777778 (3.449728) | 3.407186 (4.495186)
  12 months after trial enrollment: number analyzed (Participants) | 143 | 138
  12 months after trial enrollment | 2.377622 (3.116978) | 2.550725 (3.60266)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.1544491, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -0.6294078, 95% CI 2-sided [-1.496923 to 0.238107], Standard Error of Mean 0.4409795
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.1793486, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -0.6081765, 95% CI 2-sided [-1.497352 to 0.2809987], Standard Error of Mean 0.451915
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.6674618, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -0.1731023, 95% CI 2-sided [-0.9653829 to 0.6191784], Standard Error of Mean 0.4024787
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.5992113, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -0.2208031, 95% CI 2-sided [-1.047063 to 0.6054567], Standard Error of Mean 0.4196435

15. Secondary Outcome: Times Eating Out in the Past 7 Days
Description: Patient-reported measure of diet improvement: Number of times in the last 7 days when the patient ate fast food, takeout, or at a restaurant.
Time Frame: 6 and 12 months after trial enrollment
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: # times
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 164 | 171
# times
  6 months after trial enrollment | 4.5 (3.948285) | 4.017544 (3.78771)
  12 months after trial enrollment: number analyzed (Participants) | 144 | 138
  12 months after trial enrollment | 4.402778 (3.956617) | 4.413043 (3.927682)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.2549037, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 0.4824561, 95% CI 2-sided [-0.349686 to 1.314598], Standard Error of Mean 0.423027
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.4025977, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.3545817, 95% CI 2-sided [-0.4777863 to 1.186949], Standard Error of Mean 0.4230741
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.9825739, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -0.0102657, 95% CI 2-sided [-0.9346107 to 0.9140792], Standard Error of Mean 0.4695747
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.9443607, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -0.0340184, 95% CI 2-sided [-0.9928399 to 0.9248032], Standard Error of Mean 0.4869778

16. Secondary Outcome: Participants Answering "Yes" for Diet Improvement Compared to One Year Ago
Description: Patient-reported measure of diet improvement: Survey question: "Do you believe your diet has improved compared to one year ago?".
Time Frame: 6 and 12 months after trial enrollment
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 164 | 171
Participants
  6 months after trial enrollment | 153 | 132
  12 months after trial enrollment: number analyzed (Participants) | 144 | 136
  12 months after trial enrollment | 137 | 129
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.0000252, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 0.160997, 95% CI 2-sided [0.0868814 to 0.2351126], Standard Error of Mean 0.0376773
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.0000204, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.1691707, 95% CI 2-sided [0.0922183 to 0.2461232], Standard Error of Mean 0.0391132
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.9130816, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 0.0028595, 95% CI 2-sided [-0.0486635 to 0.0543825], Standard Error of Mean 0.0261733
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.5400053, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.0166325, 95% CI 2-sided [-0.0367394 to 0.0700045], Standard Error of Mean 0.0271062

17. Secondary Outcome: Mean Proportion of Diabetes Knowledge Questions Answered Correctly
Description: The proportion of questions testing patients' knowledge of how different factors contribute to blood sugar answered correctly.
Time Frame: 6 and 12 months after trial enrollment
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: proportion of questions
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 160 | 170
proportion of questions
  6 months after trial enrollment | 0.8267857 (0.1489169) | 0.7756302 (0.1472909)
  12 months after trial enrollment: number analyzed (Participants) | 143 | 137
  12 months after trial enrollment | 0.8271728 (0.1416987) | 0.8133472 (0.1444886)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.0018721, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 0.0511555, 95% CI 2-sided [0.0190582 to 0.0832528], Standard Error of Mean 0.016316
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.0106231, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.0433081, 95% CI 2-sided [0.0101555 to 0.0764607], Standard Error of Mean 0.0168497
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.4197898, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 0.0138256, 95% CI 2-sided [-0.0198584 to 0.0475096], Standard Error of Mean 0.0171112
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.2961479, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.0179852, 95% CI 2-sided [-0.0158442 to 0.0518147], Standard Error of Mean 0.0171811

18. Secondary Outcome: Engagement Index Score
Description: Survey-based index score for patient-reported positive engagement outcomes.
  Scores range from 0 to 1. Scores are standardized so that the control group always has a mean score of 0 and standard deviation of 1. Higher scores reflect better outcomes---here, better engagement with the program. Scores composite results from multiple survey questions while adjusting for covariance between questions.
Time Frame: 6 and 12 months after trial enrollment
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 164 | 171
score on a scale
  6 months after trial enrollment | 0.4018523 (0.8282961) | 0 (1)
  12 months after trial enrollment: number analyzed (Participants) | 144 | 138
  12 months after trial enrollment | 0.000623 (0.8280342) | 0 (1)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.0000743, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 0.4018522, 95% CI 2-sided [0.2048311 to 0.5988733], Standard Error of Mean 0.1001575
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.0004471, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.3643095, 95% CI 2-sided [0.16227 to 0.566349], Standard Error of Mean 0.1026922
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.9954683, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 0.0006229, 95% CI 2-sided [-0.2150785 to 0.2163243], Standard Error of Mean 0.1095781
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.8852268, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -0.0161147, 95% CI 2-sided [-0.2357129 to 0.2034834], Standard Error of Mean 0.1115322

19. Secondary Outcome: Number of Outpatient Visits Claimed by Insurance
Description: Healthcare utilization: Number of outpatient claims among continuously enrolled/insured subjects during the relevant time frame after trial enrollment.
Time Frame: 6 and 12 months after trial enrollment
Population: Number of participants analyzed may differ due to differences in the number of participants who remained continuously enrolled in the health plan between 6 and 12 months after trial enrollment.
Measure: Mean (Standard Deviation); unit: Number of claims
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 230 | 235
Number of claims
  6 months after trial enrollment | 5.765217 (4.884394) | 4.86383 (4.628804)
  12 months after trial enrollment | 10.1 (8.088674) | 10.07234 (8.314793)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.0417413, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 0.9013876, 95% CI 2-sided [0.0338441 to 1.768931], Standard Error of Mean 0.4414753
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.0222222, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.8939751, 95% CI 2-sided [0.1282798 to 1.65967], Standard Error of Mean 0.3896126
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.9710103, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 0.0276596, 95% CI 2-sided [-1.467185 to 1.522504], Standard Error of Mean 0.7606961
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.9539117, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.0377244, 95% CI 2-sided [-1.244338 to 1.319787], Standard Error of Mean 0.6523585

20. Secondary Outcome: Number of Inpatient and Emergency Department Visits Claimed by Insurance
Description: Healthcare utilization: Number of inpatient and emergency department claims among continuously enrolled/insured subjects during the relevant time frame after enrollment.
Time Frame: 6 and 12 months after trial enrollment
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Number of claims
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 230 | 235
Number of claims
  6 months after trial enrollment | 0.6869565 (1.363051) | 0.7914894 (1.680434)
  12 months after trial enrollment | 1.221739 (2.116365) | 1.497872 (3.350436)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.4612408, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -0.1045328, 95% CI 2-sided [-0.3830955 to 0.1740299], Standard Error of Mean 0.1417549
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.6401864, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -0.0552724, 95% CI 2-sided [-0.2874987 to 0.176954], Standard Error of Mean 0.1181649
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.2874913, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -0.2761332, 95% CI 2-sided [-0.7857084 to 0.2334419], Standard Error of Mean 0.2593125
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.4568601, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -0.155843, 95% CI 2-sided [-0.56713 to 0.2554439], Standard Error of Mean 0.2092772

21. Secondary Outcome: Proportion of Participants Filing Outpatient Insurance Claims With Insurance
Description: The number of subjects who were continuously enrolled/insured who had any outpatient claims during the relevant time frame after trial enrollment. For statistical analyses, coefficients and errors represent proportions of participants, relative to the size of the group/treatment arm.
Time Frame: 6 and 12 months after trial enrollment
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 230 | 235
Participants
  6 months after trial enrollment | 215 | 207
  12 months after trial enrollment | 221 | 224
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.0442418, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 0.0539315, 95% CI 2-sided [0.0013953 to 0.1064678], Standard Error of Mean 0.0267347
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.0454857, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.0546574, 95% CI 2-sided [0.0011025 to 0.1082124], Standard Error of Mean 0.0272506
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.683764, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 0.0076781, 95% CI 2-sided [-0.0293401 to 0.0446963], Standard Error of Mean 0.0188378
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.7708852, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.0053342, 95% CI 2-sided [-0.0306419 to 0.0413103], Standard Error of Mean 0.0183059

22. Secondary Outcome: Proportion of Participants Filing Inpatient or Emergency Department Claims With Insurance
Description: The number of subjects who were continuously enrolled/insured who had any inpatient or emergency department claims during the relevant time frame after trial enrollment. For statistical analyses, coefficients and errors represent proportions of participants, relative to the size of the group/treatment arm.
Time Frame: 6 and 12 months after trial enrollment
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 230 | 235
Participants
  6 months after trial enrollment | 70 | 84
  12 months after trial enrollment | 96 | 110
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.2245167, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -0.053099, 95% CI 2-sided [-0.1388926 to 0.0326946], Standard Error of Mean 0.0436586
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.0551913, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -0.0815933, 95% CI 2-sided [-0.1650069 to 0.0018204], Standard Error of Mean 0.0424438
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.2721373, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -0.0506938, 95% CI 2-sided [-0.1413002 to 0.0399126], Standard Error of Mean 0.0461078
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.0640071, Regression, Linear — [p-value comment as in outcome 5, analysis 2]; Mean Difference (Net) = -0.079563, 95% CI 2-sided [-0.1637776 to 0.0046516], Standard Error of Mean 0.0428514

23. Secondary Outcome: Inpatient and Emergency Department Payments
Description: Healthcare utilization: Total value (USD) of inpatient and emergency department payments among continuously enrolled/insured subjects during the relevant time frame after enrollment.
Time Frame: 6 and 12 months after trial enrollment
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: USD
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 105 | 96
USD
  6 months after trial enrollment | 2175.39 (6176.236) | 2161.593 (5284.944)
  12 months after trial enrollment: number analyzed (Participants) | 93 | 90
  12 months after trial enrollment | 3284.667 (7850.193) | 4545.119 (9951.439)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.9864081, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 13.79692, 95% CI 2-sided [-1581.244 to 1608.838], Standard Error of Mean 808.862
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.8929133, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 119.3302, 95% CI 2-sided [-1627.128 to 1865.789], Standard Error of Mean 885.2058
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.343724, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -1260.452, 95% CI 2-sided [-3880.298 to 1359.393], Standard Error of Mean 1327.743
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.3709654, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -1206.216, 95% CI 2-sided [-3860.887 to 1448.455], Standard Error of Mean 1344.574

24. Secondary Outcome: Outpatient Payments
Description: Healthcare utilization: Value (USD) of outpatient payments among continuously enrolled/insured subjects during the relevant time frame after enrollment.
Time Frame: 6 and 12 months after trial enrollment
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: USD
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 105 | 96
USD
  6 months after trial enrollment | 3313.627 (6553.01) | 2023.022 (3492.728)
  12 months after trial enrollment: number analyzed (Participants) | 93 | 90
  12 months after trial enrollment | 5327.305 (7561.854) | 4117.954 (5205.939)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.0795087, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 1290.605, 95% CI 2-sided [-153.3215 to 2734.532], Standard Error of Mean 732.2306
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.1689786, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 1207.762, 95% CI 2-sided [-517.7854 to 2933.309], Standard Error of Mean 874.6068
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.2080145, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 1209.35, 95% CI 2-sided [-679.1596 to 3097.86], Standard Error of Mean 957.1006
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.2445904, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 1258.587, 95% CI 2-sided [-869.3893 to 3386.563], Standard Error of Mean 1077.807

25. Secondary Outcome: Number of Visits to a Dietician
Description: The number of times an individual participant completed a medical appointment with a dietician in the relevant time frame, based on electronic health records.
Time Frame: 6 and 12 months after trial enrollment
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 230 | 235
number of visits
  6 months after trial enrollment | 2.656522 (1.745694) | 0.6212766 (1.263041)
  12 months after trial enrollment | 4.53913 (3.029079) | 2.919149 (2.701269)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p < 0.001, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 2.035245, 95% CI 2-sided [1.757075 to 2.313415], Standard Error of Mean 0.1415551
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p < 0.001, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 2.0087, 95% CI 2-sided [1.734473 to 2.282927], Standard Error of Mean 0.1395364
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p < 0.001, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 1.619982, 95% CI 2-sided [1.096575 to 2.143388], Standard Error of Mean 0.2663507
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p < 0.001, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 1.559642, 95% CI 2-sided [1.032797 to 2.086488], Standard Error of Mean 0.2680774

26. Secondary Outcome: Number of Diabetes Self-Management Trainings Completed
Description: The number of times an individual participant completed a Diabetes Self-Management Training (DSMT) in the relevant time frame, based on electronic health records.
Time Frame: 6 and 12 months after trial enrollment
Measure: Mean (Standard Deviation); unit: number of trainings
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 230 | 235
number of trainings
  6 months after trial enrollment | 2.243478 (1.439258) | 0.3617021 (0.7168763)
  12 months after trial enrollment | 3.791304 (2.498893) | 2.140425 (1.888297)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p < 0.001, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 1.881776, 95% CI 2-sided [1.673875 to 2.089677], Standard Error of Mean 0.1057965
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p < 0.001, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 1.868221, 95% CI 2-sided [1.664499 to 2.071943], Standard Error of Mean 0.1036609
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p < 0.001, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 1.650879, 95% CI 2-sided [1.246611 to 2.055147], Standard Error of Mean 0.2057239
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p < 0.001, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 1.636306, 95% CI 2-sided [1.232994 to 2.039618], Standard Error of Mean 0.2052192

27. Secondary Outcome: Number of Visits to an Endocrinologist
Description: The number of times an individual participant completed a medical appointment with an endocrinologist in the relevant time frame, based on electronic health records.
Time Frame: 6 and 12 months after trial enrollment
Measure: Mean (Standard Deviation); unit: number of appointments
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 230 | 235
number of appointments
  6 months after trial enrollment | 0.5913044 (0.8605437) | 0.4808511 (0.7970668)
  12 months after trial enrollment | 1.095652 (1.468588) | 0.8893617 (1.302731)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.1519153, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 0.1104533, 95% CI 2-sided [-0.040785 to 0.2616915], Standard Error of Mean 0.0769621
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.3641254, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.0594575, 95% CI 2-sided [-0.0691675 to 0.1880824], Standard Error of Mean 0.0654489
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.1100186, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = 0.2062905, 95% CI 2-sided [-0.0468859 to 0.4594669], Standard Error of Mean 0.1288363
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.2531303, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.1162375, 95% CI 2-sided [-0.0834025 to 0.3158775], Standard Error of Mean 0.1015839

28. Secondary Outcome: Number of Weight Loss and Weight Management Appointments Completed
Description: The number of times an individual participant completed a medical appointment regarding weight loss or weight management in the relevant time frame, based on electronic health records.
Time Frame: 6 and 12 months after trial enrollment
Measure: Mean (Standard Error); unit: number of appointments
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
Number analyzed (Participants) | 230 | 235
number of appointments
  6 months after trial enrollment | 0.0521739 (0.3457409) | 0.1106383 (0.5193825)
  12 months after trial enrollment | 0.0521739 (0.3457409) | 0.2212766 (0.9707113)
Statistical Analysis 1: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 6 months after trial enrollment; Test type: Superiority; p = 0.152918, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -0.0584644, 95% CI 2-sided [-0.1387132 to 0.0217844], Standard Error of Mean 0.040837
Statistical Analysis 2: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 6 months after trial enrollment; Test type: Superiority; p = 0.0548344, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -0.0585771, 95% CI 2-sided [-0.1183728 to 0.0012186], Standard Error of Mean 0.0304262
Statistical Analysis 3: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Unadjusted mean difference, 12 months after trial enrollment; Test type: Superiority; p = 0.0123238, t-test, 2 sided — Unadjusted mean difference; threshold for statistical significance: 0.05. Heteroskedasticity-robust standard errors; Mean Difference (Net) = -0.1691027, 95% CI 2-sided [-0.3013583 to -0.036847], Standard Error of Mean 0.0673022
Statistical Analysis 4: Comparison: Treatment Group-Begin Now vs Control Group-Begin Later; Adjusted mean difference for full controls, 12 months after trial enrollment; Test type: Superiority; p = 0.0032534, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -0.1701425, 95% CI 2-sided [-0.2831584 to -0.0571266], Standard Error of Mean 0.0575065

29. Other Pre Specified Outcome: Healthy Behaviors Observed in Electronic Health Record
Description: Healthy behaviors observed in electronic health record, including preventive care and appointments kept
Time Frame: 6 months and 12 months
Reporting Status: Not Posted, anticipated posting 2027-01

30. Other Pre Specified Outcome: Healthy Behaviors Observed in Paid Claims HEDIS Measures
Description: Healthy behaviors observed in paid claims using Healthcare Effectiveness Data and Information Set (HEDIS) measures. These measures were not collected for this study.
Time Frame: 6 months and 12 months
Reporting Status: Not Posted, anticipated posting 2027-01

31. Other Pre Specified Outcome: HbA1c for Household Members
Description: HbA1c available in EHR records
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Weight for Household Members
Description: Weight in pounds as available in EHR records
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

33. Other Pre Specified Outcome: BMI for Household Members
Description: BMI in kg/m^2 in pounds as available in EHR records
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Cholesterol for Household Members
Description: Cholesterol as available in EHR records
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Blood Pressure for Household Members
Description: Blood pressure as available in EHR records
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Triglycerides for Household Members
Description: Triglycerides as available in EHR records
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Fasting Glucose for Household Members
Description: Fasting glucose as available in EHR records
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Inpatient Utilization for Household Members in EHR Records
Description: Inpatient utilization for household members as available in EHR records
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

39. Other Pre Specified Outcome: Outpatient Utilization for Household Members in EHR Records
Description: Outpatient utilization for household members as available in EHR records
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

40. Other Pre Specified Outcome: Inpatient Utilization for Household Members in Paid Claims
Description: Inpatient utilization for household members as available in paid claims
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

41. Other Pre Specified Outcome: Outpatient Utilization for Household Members in Paid Claims
Description: Outpatient utilization for household members as available in paid claims
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

42. Other Pre Specified Outcome: Heterogeneity: HbA1c by Baseline Level of HbA1c
Description: Separate results by tercile of baseline HbA1c
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

43. Other Pre Specified Outcome: Heterogeneity: HbA1c by Site
Description: Heterogeneity analysis by site of the clinic
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

44. Other Pre Specified Outcome: Heterogeneity: HbA1c by Causal Tree
Description: Heterogeneity analysis by causal trees using the baseline characteristics to explore heterogeneity, sample size permitting.
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 18 months.
Description: Study was deemed minimal risk by the Institutional Review Board, and study-related adverse events and unanticipated problems were tracked.
Arm/Group | Treatment Group-Begin Now | Control Group-Begin Later
All-Cause Mortality (participants affected / at risk) | 0/249 | 0/251
Serious Adverse Events (participants affected / at risk) | 0/249 | 0/251
Other Adverse Events (participants affected / at risk) | 0/249 | 0/251

LIMITATIONS AND CAVEATS:
1. Pandemic timeperiod: Estimates were similar, though modestly powered, using only pre-pandemic data.
2. Effects may differ at other health systems / patients who are not well connect to a system.
3. Wait list design: control group members may take additional actions due to awareness of the program.
4. Lack of detailed recall measures.
5. It may take longer than 6-12 months for the intervention to change these outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/32/NCT03718832/Prot_001.pdf
  • Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT03718832/SAP_000.pdf